CLINICAL TRIAL: NCT02791217
Title: Identification of Hematological Malignancies and Therapy Predication Using microRNAs as a Diagnostic Tool
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assuta Medical Center (Other)
Collaborators: Laniado Hospital (Other)
Responsible Party: Principal Investigator, shpilberg ofer, Head of hematology department, Assuta Medical Center
Other Study IDs: 2015097
Record Dates: First submitted 2016-05-30; First posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Lymphoma, B-Cell; Follicular Lymphoma; Hodgkin Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Follicular; Hodgkin Disease; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Diffused Large B cell Lymphoma
- Follicular Lymphoma
- Multiple Myeloma
- Hodgkin Lymphoma
- Healthy individuals

SUMMARY:
MiRNAs are small (~19-25 nucleotides) non-coding RNA molecules that bind to mRNA in a sequence-specific manner. MiRNAs regulate gene expression at the post-transcriptional level. MiRNAs regulate critical cell processes such as metabolism, apoptosis, development, cell cycle, hematopoietic differentiation and have been implicated in the development and progression of several types of cancers, including hematological malignancies. Over-expression, amplification and/or deletion of miRNAs and miRNA-mediated modification of epigenetic silencing can all lead to oncogenic pathways.

Hematologic cancers, which are caused by the malignant transformation of bone marrow cells and the lymphatic system, are usually divided into three major clusters: leukemia, lymphoma, and multiple myeloma. To date, some of the hematological malignancies are very aggressive that early diagnosis is essential for improving prognosis and increasing survival rates. However, current diagnostic methods have various limitations, such as insufficient sensitivity, specificity, it is also time-consuming, costly, and requires a high level of expertise, which limits its application in clinical contexts. Thus, development of new biomarkers for the early detection and relapse of hematological malignancies is desirable.

Some of the innate properties of miRNAs make them highly attractive as potential biomarkers. MiRNAs can be readily detected in small volume samples using specific and sensitive quantitative real-time PCR; they have been isolated from most body fluids, including serum, plasma, urine, saliva, tears and semen and are known to circulate in a highly stable, cell-free form. They are highly conserved between species, allowing the use of animal models of disease for pre-clinical studies. Furthermore, tumor cells have been shown to release miRNAs into the circulation and profiles of miRNAs are altered in the plasma and/or serum of patients with cancer. A growing number of publications confirm that miRNAs can be a useful biomarker for hematological malignancies diagnosis and progression.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnose patients with: Diffused large B cell lymphoma, Follicular lymphoma, Multiple myeloma and Hodgkin lymphoma.
* Patients after chemotherapy (5-30 days).
* Above age 18.

Exclusion Criteria:

* Non-HIV/HCV/HBV Below age 18.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diffused Large B cell Lymphoma Follicular Lymphoma Multiple Myeloma Hodgkin Lymphoma Healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Molecular characteristics (by GEP, miRNA) | 1 year

SECONDARY OUTCOMES:
Event free survival (EFS) | 0-5 years
Overall survival (OS) | 0-5 years

IPD SHARING:
Plan to Share IPD: Undecided